CLINICAL TRIAL: NCT02362750
Title: Evaluating Cancer Survivorship Care Models
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: IH-12-11-5255
Record Dates: First submitted 2015-01-21; First posted 2015-02-13 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Quality of Life; Cancer
Keywords: comparative effectiveness; survivorship; Patient-Centered Outcomes Research
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Participating Program Administrators: Eligible survivorship program administrators at selected Commission on Cancer-accredited institutions will complete an organizational interview and organizational survey.
  Interventions: Other: Organizational Interview; Other: Organizational Survey
- Participating Cancer Survivors: Survivors receiving follow-up care surveys at selected Commission on Cancer-accredited institutions will complete four surveys:
  Survivor Survey (1): Pre-Visit Baseline Survivor Survey (2): 1 Week Post-Visit Survivor Survey (3): 3 Months Post-Visit Survivor Survey (4): 6 Months Post-Visit
  Interventions: Other: Survivor Survey (1): Pre-Visit Baseline; Other: Survivor Survey (2): Post-Visit; Other: Survivor Survey (3): 3 Month Post-Visit; Other: Survivor Survey (4): 6 Month Post-Visit
- Participating Clinicians: Survivorship clinicians from clinical survivorship programs at selected Commission on Cancer-accredited institutions will complete a clinician survey.
  Interventions: Other: Clinician Survey

INTERVENTIONS:
Other: Organizational Interview — Survivorship program leaders will participate in a phone-based organizational interview regarding the organization of the clinical survivorship care program.
  Groups: Participating Program Administrators
Other: Organizational Survey — Survivorship program leaders will participate in a brief web-based organizational survey regarding the organization of the clinical survivorship care program.
  Groups: Participating Program Administrators
Other: Survivor Survey (1): Pre-Visit Baseline — Survivors will participate in a baseline survey regarding their satisfaction, health-related quality of life, ability to manage their cancer post-treatment and appropriate health care utilization.
  Groups: Participating Cancer Survivors
Other: Survivor Survey (2): Post-Visit — Survivors will participate in a survey within one week after their survivorship visit regarding their satisfaction, health-related quality of life, ability to manage their cancer post-treatment and appropriate health care utilization.
  Groups: Participating Cancer Survivors
Other: Survivor Survey (3): 3 Month Post-Visit — Survivors will participate in a survey three months after their survivorship visit regarding their satisfaction, health-related quality of life, ability to manage their cancer post-treatment and appropriate health care utilization.
  Groups: Participating Cancer Survivors
Other: Survivor Survey (4): 6 Month Post-Visit — Survivors will participate in a survey six months after their survivorship visit regarding their satisfaction, health-related quality of life, ability to manage their cancer post-treatment and appropriate health care utilization.
  Groups: Participating Cancer Survivors
Other: Clinician Survey — Survivorship program clinicians will complete a survey for each survivor who enrolls in the study indicating services provided through the survivorship visit.
  Groups: Participating Clinicians

SUMMARY:
The Evaluating Cancer Survivorship Care Models project is an innovative 3-year study that is collecting data to help understand how to best deliver follow-up care to cancer survivors. Cancer is a complex disease requiring complex treatments that can cause lasting impacts after treatment ends. Some patients face physical, psychosocial, spiritual and/or practical challenges as they adjust to life after cancer. Fortunately, health care providers have begun to focus on the consequences of cancer and its treatment and are more actively working with cancer survivors to manage post-treatment needs and care.

Led by the George Washington University and funded by the Patient-Centered Outcomes Research Institute, this project brings together representatives from the Commission on Cancer, the Cancer Support Community, LIVESTRONG and the American Cancer Society as well as cancer survivors and healthcare professionals to better understand how different strategies or models of care impact outcomes that are most important to cancer survivors. The project will focus on survivors of breast, prostate and colorectal cancers and will be relevant for understanding the needs and preferences of survivors of other cancers as well. The emphasis is on patient-centered outcomes, which are outcomes that are most significant to patients, such as patient satisfaction and quality of life.

DETAILED DESCRIPTION:
Evaluating Cancer Survivorship Care Models Study Overview and Research Design

Cancer is a complex disease requiring complex treatments that can cause lasting impacts after treatment ends. Some patients face lasting physical, psychosocial, spiritual and/or practical challenges as they adjust to life after cancer. Fortunately, health care clinicians have begun to focus on the consequences of cancer and its treatment and are more actively working with cancer survivors to manage post-treatment needs and care.

The Evaluating Cancer Survivorship Care Models project is a groundbreaking 3-year comparative effectiveness research (CER) study that examines how to best deliver follow-up care to cancer survivors. This project is led by the George Washington University and funded by the Patient-Centered Outcomes Research Institute. A key component of the project is the use of a stakeholder Advisory Board chaired by a cancer survivor who serves as a senior advisor to the research team. The Advisory Board includes survivors, survivor advocates, clinicians, health care professionals and advisors from stakeholders across myriad facets of cancer care, including the Cancer Support Community, LIVESTRONG, the Commission on Cancer, and the American Cancer Society. These organizations are critical to the success of the project.

The study is innovative in its focus on patient-centered outcomes. The first phase of the project employed a mixed methods approach including a secondary analysis of existing data from 4 national surveys, focus groups with cancer survivors, an environmental scan of existing survivorship programs and a national survey of cancer survivors to develop an outcomes tool and a prospective observational CER study. Based on results from the first phase, the study team at the George Washington University (GW) developed a patient-prioritized index to identify services and components of care that patients equate with high quality survivorship care.

Three models of survivorship care at Commission on Cancer-accredited institutions were identified through the environmental scan. In the CER phase of the study, each survivorship care model will serve as a comparator for the other two models. Patients in the CER study population will be adults who have been diagnosed with non-metastatic breast, prostate or colorectal cancer and completed active treatment. Patient-reported outcomes will be assessed at three points in the project: at baseline (immediately prior to and immediately following a post-treatment survivorship visit), 3 months post-visit and 6 months post-visit. Multivariable analyses including repeated measures and mixed-effect regression modeling will be used to control for systematic differences across the groups, which would further increase the validity of our results. Using the newly-developed index, the comparative effectiveness study will measure the quality of programs according to what patients have identified as most important to them.

The investigators have launched the CER phase of the study and are enrolling high-performing survivorship programs. Our pool of invited participants consists of Commission on Cancer-accredited sites with clinical survivorship care programs that meet the following eligibility criteria:

* Provide services to survivors of breast, prostate or colorectal cancer
* Have demonstrated a high performance level on incorporating elements of survivorship care into clinical care delivery
* See at least 60 new survivors yearly
* Includes the most common characteristics related to delivery of survivorship care

During the CER study, data will be gathered from survivorship program administrators, patients and survivorship care clinicians. Survivorship program administrators will complete an interview and survey to examine how survivorship programs are organized and identify key characteristics of programs to determine which factors are most influential in delivering high quality post-treatment survivorship care. Patients will complete surveys measuring patient-centered outcomes: health-related quality of life; self-efficacy; satisfaction; health care utilization and a newly developed measure of quality of survivorship care as prioritized by patients. Clinicians will complete surveys on the services offered during participating patients' initial post-treatment survivorship visit. Together, this data will allow the GW study team to understand successful strategies for transforming the care delivery system to be more responsive to patient needs.

In the third and final phase, this project will generate critical data for a variety of decision-makers related to care for post-treatment cancer survivors and will result in evidence-based guidance for how to organize and deliver post-treatment care. The GW study team seeks to provide recommendations on survivorship care delivery best practices; develop tools for improving survivorship programs and care delivery from both clinician and patient perspectives; and to widely disseminate findings to a variety of stakeholders, including survivors and their families, clinicians, survivorship care program leaders, payers, policymakers and others.

ELIGIBILITY:
Inclusion criteria for the CER component:

Survivorship program administrators oversee survivorship programs which:

* See at least 60 new survivors of non-metastatic breast, prostate or colorectal cancer or survivors of any type of cancer yearly
* Represent one of the clinical survivorship care models identified in our environmental scan
* Indicate a high performance level on incorporating elements of survivorship care into clinical care delivery.

Survivors:

* English-speaking survivors of non-metastatic breast, prostate or colorectal cancers
* Completed planned active treatment (chemotherapy, radiation, and/or surgery) with the exception of hormonal medication, aromatase inhibitors or other maintenance therapy
* Diagnosed at 18 years old or older
* First appointment with the survivorship program is planned but has not yet been completed

Survivorship program clinicians:

• Must be providing services for eligible survivors who have completed their first visit with the survivorship program and are participating in the study.

Exclusion criteria for the CER component:

Survivorship program administrators:

* Programs with fewer than at least 60 new survivors yearly
* Do not provide services to adult survivors of non-metastatic breast, prostate or colorectal cancer or survivors of any type of cancer
* Do not represent one of the three models of clinical survivorship care as identified in our environmental scan
* Do not indicate a high performance level on incorporating elements of survivorship care into clinical care delivery

Survivors:

* Received diagnosis for cancer that was not breast, prostate or colorectal cancer
* Not English-speaking
* Currently undergoing active treatment (defined as chemotherapy, radiation, and/or surgery)
* Cancer has metastasized
* Diagnosed at under 18 years old
* Have completed first appointment with the survivorship program

Men will be excluded from the breast cancer arm of the study. Women will be excluded from the prostate cancer arm of the study.

Survivorship program clinicians:

• Not providing services for eligible survivors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1 of our study focused on developing instruments to conduct comparative effectiveness research. The investigators analyzed three large national studies of cancer survivors; conducted focus groups across the country with adult survivors of breast, prostate or colorectal cancer; surveyed Commission on Cancer accredited institutions regarding provision of survivorship care and surveyed a nationally representative sample of adult cancer survivors. In phase II, the investigators will conduct surveys with survivorship program leaders at eligible Commission on Cancer accredited institutions; adult survivors of breast, prostate or colorectal cancer; and the survivorship program clinicians providing their care.
Sampling Method: Non-Probability Sample
Enrollment: 992 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Patient-centered outcomes for cancer survivors | Patients will be surveyed before their survivorship visit, within 1 week after survivorship visit, 3 months after survivorship visit and 6 months after survivorship visit
  The investigators will assess the following specific outcomes across different cancer survivorship care models for the comparative effectiveness evaluation: a Patient Index and patients' satisfaction, health-related quality of life, ability to manage their cancer post-treatment and appropriate health care utilization. Each cancer survivorship care model identified through the study will serve as a comparator for the other two models.

CONTACTS AND LOCATIONS:
Overall Officials: K. Holly Mead, PhD, Principal Investigator — The George Washington University
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Mead KH, Wang Y, Cleary S, Arem H, Pratt-Chapman ML. Defining a patient-centered approach to cancer survivorship care: development of the patient centered survivorship care index (PC-SCI). BMC Health Serv Res. 2021 Dec 18;21(1):1353. doi: 10.1186/s12913-021-07356-6. PMID 34922530
- See also: American Cancer Society. Cancer Treatment and Survivorship Facts & Figures 2012-2013. Atlanta: American Cancer Society; 2012. — http://www.cancer.org/acs/groups/content/@epidemiologysurveilance/documents/document/acspc-033876.pdf
- See also: Viswanathan M, Halpern M, Swinson Evans T, et al. Models of Cancer Survivorship Care [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2014 Mar. (Technical Briefs, No. 14.) — http://www.ncbi.nlm.nih.gov/books/NBK196214/